CLINICAL TRIAL: NCT05217862
Title: The Implications of Not Imposing COVID-19 Testing on Patients Prior to Elective Cataract Surgery
Brief Title: Effect Not Imposing COVID-19 Testing Prior to Elective Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdelazeem, Associate professor of Ophthalmology, Assiut University
Other Study IDs: 17300720
Record Dates: First submitted 2022-01-29; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Cataract Surgery; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PCR for COVID-19 testing — PCR for asymptomatic adult undergoing elective cataract surgery

SUMMARY:
The world health organization declared corona virus disease (COVID19) a pandemic since march 2020. Since then the future landscape of medical practices and procedures is being heavily shaped by the emergence of this pandemic. COVID 19 testing has already standardized within the medical field as doctors wearing scrubs or fitness examination before operation. We are now more than 2 years into COVID-19 pandemic with more than 6 effective vaccines available in the market for public to boost and build up their immunity against the virus. Every 3 to 4 months we hear about a new strain and another wave of the virus attacking the world, therefore healthcare institutions face enormous challenges in balancing patients' needs and simultaneous safety to health care workers.

The Indian council of medical research in June 2020 proposed that testing for Covid-19 for asymptomatic patients coming for elective surgeries should be performed for neurosurgery, ear nose, and throat (ENT) surgery, dental procedures, etc. and for non-surgical interventions like bronchoscopy, upper gastrointestinal endoscopy and dialysis. A role of preoperative testing of Covid-19 for every patient is still controversial especially in asymptomatic healthy patients with not known exposure to a COVID positive patient.

Most patients attending eye out patient department (EOPD) are aged 65y and older are considered at a higher risk for worse outcome in case of COVID-19 infection. Therefore a rethink of a cataract surgery pathway should include preoperative perioperative and postoperative care in order to maintain safety conditions for patients and for healthcare staff.

COVID-19 can infect anyone and result in transmission of infection before the patient become symptomatic or even without ever developing symptoms. Therefore preoperative screening of patients undergoing ophthalmic surgery should be considered.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic adult undergoing cataract surgery

Exclusion Criteria:

* Symptomatic patients (fever, cough lethargy malaise , headache, and aches, sore throat and diarrhoea

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asymptomatic adult undergoing cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-01-29 (Actual)

PRIMARY OUTCOMES:
To identify +ve or -ve COVID patient | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt